CLINICAL TRIAL: NCT06119295
Title: Investigating the Effects of Altering Portion Size Reduction Awareness on Compensatory Eating Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Portion size reduction study
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2023-11

CONDITIONS: Eating Behavior; Obesity
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Condition (Experimental): Participants will be served a lunch - this will be of a fixed portion - this portion size will be the same amount of food as was consumed in the ad libitum lunch meal in the baseline session (participants will be told that the amount of food served is the same as the amount they consumed in the baseline session).
  Interventions: Behavioral: Portion size manipulation
- Reduce aware condition (Experimental): Participants will be served a lunch - this will be of a fixed portion - this portion size will be 15% less than the amount of food consumed in the ad libitum lunch meal in the baseline session (participants will be told that the amount of food served has been reduced from the amount they consumed in the baseline session).
  Interventions: Behavioral: Portion size manipulation
- Reduced unaware condition (Experimental): Participants will be served a lunch - this will be of a fixed portion - this portion size will be 15% less than the amount of food consumed in the ad libitum lunch meal in the baseline session (participants will be told that the amount of food served is the same as the amount they consumed in the baseline session).
  Interventions: Behavioral: Portion size manipulation

INTERVENTIONS:
Behavioral: Portion size manipulation — The intervention will be administered via changing portion sizes of foods served to participants. Depending on the condition participants are in, they will be served either a portion size which consists of the amount of food they consumed in the first test session, or a reduced portion size. Within these two reduced portion size conditions, one group of participants will be made aware that their portion size has been reduced, the other will not and instead will be told that this portion size is the same as the amount of food they consumed in the previous session.

SUMMARY:
The present study aims to investigate whether energy intake is reduced when participants consume a reduced portion size (15% compared to the 'control' portion), and also to see whether awareness of this reduction affects energy intake.

DETAILED DESCRIPTION:
In the present study, all participants will participate in two sessions - the baseline session and the experimental session. In the baseline session, participants will be given ad libitum access to a lunch meal (followed by ad libitum access to dessert), and ad libitum access to a dinner meal (followed by ad libitum access to dessert). Then, after a washout period of between 1-6 weeks, participants will return to complete the experimental session, where they will be randomised to one of three conditions:

Condition 1 (control condition): The same as the baseline condition except that the lunch will be of a fixed portion which participants must consume all of - this portion size will be the same amount of food as was consumed in the ad libitum lunch meal in the baseline session (participants will be told that the amount of food served is the same as the amount they consumed in the baseline session).

Condition 2 (reduced aware condition): The same as the baseline condition except that the lunch will be of a fixed portion which participants must consume all of - this portion size will be 15% less than the amount of food consumed in the ad libitum lunch meal in the baseline session (participants will be told that the amount of food served has been reduced from the amount they consumed in the baseline session).

Condition 3 (reduced unaware condition): The same as the baseline condition except that the lunch will be of a fixed portion which participants must consume all of - this portion size will be 15% less than the amount of food consumed in the ad libitum lunch meal in the baseline session (participants will be told that the amount of food served is the same as the amount they consumed in the baseline session).

ELIGIBILITY:
Inclusion Criteria:

* United Kingdom (UK) residents able to visit laboratory on campus in Liverpool, aged ≥ 18
* Body Mass Index (BMI) between 18.5 and 32.5 kg/m2
* Proficiency in English language
* Self-report willingness to eat each of the test foods

Exclusion Criteria:

* Current medication use which affects appetite
* Pregnant
* Currently or previously diagnosed with an eating disorder
* Currently on a diet
* Have any food allergies or intolerances
* Are vegan

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Immediate energy intake post-fixed lunch meal | Within 30 minutes after intervention administered
  Amount of energy consumed from the lunch dessert
Total delayed post-fixed lunch meal energy intake | Within 10 hours after intervention administered
  Amount of energy consumed from the post-lunch snack box intake, dinner meal, dinner dessert, post-dinner snack box intake, additional energy intake
Total post-fixed lunch meal energy intake | Within 10 hours after intervention administered
  Amount of energy consumed from the lunch dessert, post-lunch snack box intake, dinner meal, dinner dessert, post-dinner snack box intake, additional energy intake

SECONDARY OUTCOMES:
Post-lunch snack box intake | Within 4 hours after intervention administered
  Amount of energy consumed from snack box consumed between lunch and dinner
Total intake of the ad libitum dinner meal | Within 4-5 hours after intervention administered
  Amount of energy consumed from the dinner meal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised data set will be published on the open science framework for anyone to access.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available after data collection has finished, this will be available indefinitely.